CLINICAL TRIAL: NCT00322894
Title: Expanded Breast Cancer Registry and Tissue Repository
Status: Completed | Type: Observational
Sponsor: New Mexico Cancer Research Alliance (Other)
Collaborators: University of New Mexico (Other)
Responsible Party: Sponsor
Other Study IDs: INST 0552C
Record Dates: First submitted 2006-05-05; First posted 2006-05-08 (Estimated); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Risk factors; Treatment; Clinico-pathologic; Outcomes; Tissue repository; Registry
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Biospecimen Retention: Samples With DNA — Sample of tumor, buccal cells and blood collected at the time of study enrollment.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The Expanded Breast Cancer Registry and Tissue Repository Research Team (EBCR-RT) is comprised of University of Mexico Comprehensive Cancer Center faculty and staff whose goals are to improve the outcomes and quality of life of patients with breast cancer, and ultimately to eradicate and cure breast cancer. One focus of the EBCR-RT is the creation an infrastructure that can potentially be adopted as a model for a statewide registry and tissue repository for the discovery of biomarkers for this disease.

The goals of the EBCR are:

1. To register patients diagnosed with breast cancer and information relevant to their diagnosis (such as stage, grade, hormone receptor status, etc), treatment (surgery, radiation, chemotherapy, hormone therapy, etc), and survivorship (Quallity of Life, etc).
2. To collect relevant demographics including age, menopausal status, race/ethnicity, body mass index (BMI), place of residence, behaviors (smoking, alcohol intake, etc)
3. To establish a paired tumor tissue and blood sample for each relevant time-point (as defined in the protocol), which will be stored in the Tissue Bank Shared Resource Facility for future hypothesis-driven research.

DETAILED DESCRIPTION:
Institutions and/or physicians are required to report each new diagnosis of breast cancer to the New Mexico Tumor Registry (NMTR). The NMTR is a valuable database that provides information on breast cancer, including trends in incidence and survival. However, relevant information on breast cancer prognosis and treatment is either not routinely collected or not readily available to the NMTR. We propose to establish an Expanded Breast Cancer Registry and Tissue Repository (EBCR) at this institution that could serve as an infrastructure for collection of this information. Furthermore, a tissue bank will be established for collection of paired tissue (tumor, buccal cells and blood sample) from patients diagnosed with breast cancer who consent to providing excess/extra tissue and additional blood for the Tissue Repository. This tissue bank will serve as a repository from which researchers can access tissue samples to conduct laboratory-based studies of genetic determinants of breast cancer risks, prognosis and survival in women with breast cancer seen in this institution.

ELIGIBILITY:
Inclusion Criteria:

* All patients diagnosed with breast cancer, regardless of gender, ethnicity/race, stage of disease or treatment, are eligible.
* Patients must be less than or equal to one year from diagnosis of non-metastatic breast cancer OR less than or equal to one year from initiation of treatment for metastatic disease.
* Pathological diagnosis of breast cancer
* Expected availability of clinical follow up data
* Eighteen years old or older
* Participants must be willing to provide written, informed consent obtained in accordance with institutional and federal guidelines

Exclusion Criteria:

* Not specified.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients diagnosed with breast cancer during the study period commencing January 2006, regardless of gender, ethnicity/race, stage of disease or treatment.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2006-02-16 (Actual); Primary Completion 2016-08-02 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Identify risk factors for breast cancer | 4 years
  Prospectively collect demographic, risk factor, diagnosis and treatment data and tissues (blood, buccal cells and tumor if appicable) for breast cancer patients seen at the UNM Cancer Center to assist in identification of unique factors that may impact patient prognosis in this population.

SECONDARY OUTCOMES:
Establish a centralized tissue repository | 4 years
  Establish a centralized tissue repository (breast and related tissues) to serve as a resource for current and future scientific studies.

OTHER OUTCOMES:
Assess clinico-pathologiv variables and outcomes | 10 years
  Utilize the Extended Breast Cancer Repository clinical database to determine the relationship between clinico-pathologic variables and patient outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Royce, MD, Principal Investigator — University of New Mexico Cancer Center
Locations (1):
- University of New Mexico Comprehensive Cancer Center, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: University of New Mexico Cancer Center — http://www.cancer.unm.edu
- See also: New Mexico Cancer Care Alliance — http://www.nmcca.org